CLINICAL TRIAL: NCT04945798
Title: Effects of Osteopathic Manipulative Treatment of Fascial Restrictions on Body Awareness, Mood, and Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BHS1611
Record Dates: First submitted 2021-03-10; First posted 2021-06-30 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Segmental and Somatic Dysfunction of Other Regions (M99.09)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No OMT (No Intervention): The STAI (Y2), DASS and Scale of Body Connection administered to this cohort at baseline (T1), after two treatments (T3), and after four treatments (T4).
- OMT (Active Comparator): OMT: direct myofascial release for the triplanar diagnonosis to the OA, thoracic outlet, respiratory diaphragm and pelvic diaphragm concluding with a pedal pump for 120 seconds.
  The STAI (Y2), DASS and Scale of Body Connection administered to this cohort at baseline (T1), after two treatments (T3), and after four treatments (T4).
  Interventions: Other: OMT

INTERVENTIONS:
Other: OMT — OMT: direct myofascial release for the triplanar diagnonosis to the OA, thoracic outlet, respiratory diaphragm and pelvic diaphragm concluding with a pedal pump for 120 seconds
  Arms: OMT

SUMMARY:
The purpose of this research is to assess the effects osteopathic manipulative treatment (OMT) of fascial strain patterns on body awareness, proprioception, and mood.

ELIGIBILITY:
Inclusion Criteria:

* Functionally healthy adults that can move all four limbs within normal range of motion.

Exclusion Criteria:

* People with the following conditions may not participate in the study: known bony injuries or fractures, open wounds, abscesses, infections of the soft tissue or bones, malignancies, auto-immune disorders affecting the musculoskeletal system (ex. lupus, rheumatoid arthritis), severe osteoporosis, aortic aneurysm, deep venous thrombosis, history of pulmonary embolism, bleeding disorders, neurovascular compromise, anticoagulation therapy, recent surgery, recent herniated discs, unstable heart conditions, and musculoskeletal strains or sprains, enlarged spleen or liver, mononucleosis, pregnancy, untreated hyperthyroidism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Proprioception: Active Hip Flexion Position Detection. | 4 weeks
  Measurements use a goniometer. Measurements are in degrees. Participant judges accuracy of position on a scale of 1-5: 1= very inaccurate, 2= somewhat inaccurate, 3=neutral, 4= somewhat accurate, 5= very accurate.
Proprioception: Active Shoulder Joint Position Detection. | 4 weeks
  Measurements use a goniometer. Measurements are in degrees. Participant judges accuracy of position on a scale of 1-5: 1= very inaccurate, 2= somewhat inaccurate, 3=neutral, 4= somewhat accurate, 5= very accurate.
Proprioception: Active Thoracolumbar Position Detection. | 4 weeks
  Measurements use a goniometer. Measurements are in degrees. Participant judges accuracy of position on a scale of 1-5: 1= very inaccurate, 2= somewhat inaccurate, 3=neutral, 4= somewhat accurate, 5= very accurate.
Body Awareness: Scale of Body Connection | 4 weeks
  A higher score represents better outcomes with increased body awareness. Minimum score: 0. Maximum for whole scale: 4. Scores are based on 12 items for body awareness (BA) and 8 items for body dissociation (BD). The items are scored on a 5-point scale, ranging from 0-4 with 0 at "not at all" and 4 at "all of the time." To score the BA subscale: sum the endorsed items and divide by the total number of items (12). To score the DB subscale: sum the endorsed items and divide by the total number of items (8). A positive change on the BA scale would represent an increase in bodily awareness, and a positive result. A negative change on the DB scale would represent a decrease in bodily dissociation, and a positive result.
Mood: Depression Anxiety Stress Scale. | 4 weeks
  Increasing scores are associated with depression, anxiety, or stress. Items are scored within three subscales: depression, anxiety and stress. For individual subscales the scoring is as follows. Depression: normal (0-9), mild (10-13), moderate (14-20), severe (21-27), extremely severe (28+). Anxiety: normal (0-7), mild (8-9), moderate (10-14), severe (15-19), extremely severe (20+). Stress: normal (0-14), mild (15-18), moderate (19-25), severe (26-33), extremely severe (34+). Minimum score is 0 and maximum score is 126 for the entire scale.
Mood: State Trait Anxiety Inventory Form Y-2. | 4 weeks
  A higher score is associated with increased anxiety trait. The minimum score is 20. The maximum score is 80. The range for no or little anxiety is 20-37. Moderate anxiety scores are from 38-44. High anxiety range is from 45-80.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Suessle, DO, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology College of Osteopathic Medicine at Arkansas State University, Jonesboro, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trevithick A, Park SY. A Novel Method for Assessment of Proprioception. Journal of Emerging Investigators. 2018. https://www.emerginginvestigators.org/articles/a-novel-method-for-assessment-of-proprioception/pdf. Published June 22, 2018. Accessed January 7, 2021.
- [Background] Price CJ, Thompson EA. Measuring dimensions of body connection: body awareness and bodily dissociation. J Altern Complement Med. 2007 Nov;13(9):945-53. doi: 10.1089/acm.2007.0537. PMID 18047441
- [Background] Kosmahl EM. Goniometry: Thoraco-Lumbar Spine Sidebending. The University of Scranton. https://www.scranton.edu/faculty/kosmahl/courses/gonio/spine/pages/thor-side.shtml. Accessed February 1, 2021.
- [Background] Seffinger MA, executive ed. Foundations of Osteopathic Medicine: Philosophy, Science, Clinical Applications, and Research. 4th ed. Philadelphia, PA: Wolters Kluwer Health/Lippincott Williams & Wilkins; 2018.
- [Background] Chila AG, executive ed. Foundations of Osteopathic Medicine. 3rd ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2011.
- [Background] Beatty DR. The Pocket Manual of OMT. 2nd ed. Philadelphia, PA: Lippincott Williams & Wilkins/Wolters Kluwer Health, Inc.; 2011.
- [Background] Lovibond, S.H. & Lovibond, P.F. Manual for the Depression Anxiety Stress Scales. 2nd edition. 1995. Sydney: Psychology Foundation. http://www2.psy.unsw.edu.au/dass/Download%20files/Dass42.pdf. Updated July 26, 2018. Accessed January 23, 2021.
- [Background] Measurement of Range of Motion of the Hip. Musculoskeletal Key. https://musculoskeletalkey.com/measurement-of-range-of-motion-of-the-hip/. Published August 10, 2016. Accessed February 1, 2021.
- [Background] Nicholas AS; Nicholas EA. In: Atlas of Osteopathic Techniques. 3rd ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2016.
- [Background] Speilberger CD. State Trait Anxiety Inventory for Adults. Mind Garden, Inc. www.mindgarden.com. 1977. Accessed December 31, 2020.
- [Background] van der Wal J. The architecture of the connective tissue in the musculoskeletal system-an often overlooked functional parameter as to proprioception in the locomotor apparatus. Int J Ther Massage Bodywork. 2009 Dec 7;2(4):9-23. doi: 10.3822/ijtmb.v2i4.62. PMID 21589740